CLINICAL TRIAL: NCT03043872
Title: A Phase III, Randomized, Multicenter,Open-Label, Comparative Study to Determine the Efficacy of Durvalumab or Durvalumab and Tremelimumab in Combination With Platinum-Based Chemotherapy for the First-Line Treatment in Patients With Extensive Disease Small-Cell Lung Cancer (SCLC) (CASPIAN)
Brief Title: Durvalumab ± Tremelimumab in Combination With Platinum Based Chemotherapy in Untreated Extensive-Stage Small Cell Lung Cancer (CASPIAN)
Acronym: CASPIAN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419QC00001; 2016-001203-23 (EudraCT Number)
Record Dates: First submitted 2017-01-18; First posted 2017-02-06 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Carcinoma Extensive Disease
Keywords: Carcinoma, Small Cell Lung; Oat Cell Carcinoma of Lung; Oat Cell Lung Cancer; Small Cell Cancer Of The Lung; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; tremelimumab; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): durvalumab+tremelimumab+EP (carboplatin or cisplatin + etoposide)
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide
- Arm 2 (Experimental): durvalumab+EP (carboplatin or cisplatin + etoposide)
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide
- Arm 3 (Active Comparator): EP (carboplatin or cisplatin + etoposide)
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Durvalumab — IV infusions every 3 weeks for 12 weeks (4 cycles) and every 4 weeks thereafter until PD or other discontinuation criteria.
  Arms: Arm 1; Arm 2
Drug: Tremelimumab — IV infusions every 3 weeks for 12 weeks(4 cycles). An additional dose of tremelimumab will be administered in the week 16.
  Arms: Arm 1
Drug: Carboplatin — up to 4 cycles every 3 weeks in Arm 1 and 2, up to 6 cycles every 3 weeks in Arm 3
Drug: Cisplatin — up to 4 cycles every 3 weeks in Arm 1 and 2, up to 6 cycles every 3 weeks in Arm 3
Drug: Etoposide — up to 4 cycles every 3 weeks in Arm 1 and 2, up to 6 cycles every 3 weeks in Arm 3

SUMMARY:
This is a phase III, randomized, open-label, multicenter, global study to determine the efficacy and safety of combining durvalumab ± tremelimumab with platinum based chemotherapy (EP) followed by durvalumab ± tremelimumab maintenance therapy versus EP alone as first-line treatment in patients with extensive-stage small-cell lung cancer

DETAILED DESCRIPTION:
Primary objective of this study is to assess the efficacy of durvalumab + tremelimumab + EP treatment compared with EP and the efficacy of durvalumab + EP treatment compared with EP in terms of OS.

All patients will be randomized in a 1:1:1 ratio in a stratified manner according to the planned platinum-based therapy for Cycle 1 (cisplatin or carboplatin) to receive treatment with durvalumab + tremelimumab + EP (Arm 1), durvalumab + EP (Arm 2), or standard of care- EP (Arm 3). Arm 1 and Arm 2 patients receive the treatment until confirmed disease progression while Arm 3 patients receive up to 6 cycles of EP and prophylactic cranial irradiation if clinically indicated, at the Investigators' discretion.Patients who have discontinued treatment due to toxicity or symptomatic deterioration, clinical progression, or who have commenced subsequent anticancer therapy will be followed up until confirmed disease progression and for survival.

Targeted population are adult patients (aged ≥18 years) with histologically or cytologically documented extensive disease (American Joint Committee on Cancer Stage (7th edition) IV SCLC [T any, N any,M1 a/b]), or T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan. Patients must have WHO/ECOG performance status of 0 or 1.

Tumor assessments will be performed at Screening as baseline with follow-up at Week 6 ±1 week from the date of randomization, at Week 12 ±1 week from the date of randomization, and then every 8 weeks ±1 week until confirmed objective disease progression.

An independent data monitoring committee (IDMC) comprised of independent experts will be convened to confirm the safety and tolerability of the proposed dose and schedule of durvalumab ± tremelimumab in combination with platinum based chemotherapy at two early stages of enrolment.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically documented extensive disease. Brain metastases; must be asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment.
2. Suitable to receive a platinum-based chemotherapy regimen as 1st line treatment.
3. Life expectancy ≥12 weeks at Day 1.
4. ECOG 0 or 1 at enrolment.
5. No prior exposure to immune-mediated therapy excluding therapeutic anticancer vaccines.

Exclusion criteria:

1. Any history of radiotherapy to the chest prior to systemic therapy or planned consolidation chest radiation therapy (except paliative care outside of the chest).
2. Paraneoplastic syndrome of autoimmune nature, requiring systemic treatment or clinical symptomatology suggesting worsening of PNS
3. Active infection including tuberculosis, HIV, hepatitis B anc C
4. Active or prior documented autoimmune or inflammatory disorders
5. Uncontrolled intercurrent illness, including but not limited to interstitial lung disease.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyi Jiang, M.D., Study Director — AstraZeneca
Locations (171):
- United States (19):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Rogers, Arkansas
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Athens, Georgia
  - Research Site, Fort Wayne, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Leawood, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Paducah, Kentucky
  - Research Site, Grand Rapids, Michigan
  - Research Site, Mineola, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Nashville, Tennessee
  - Research Site, Kennewick, Washington
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Austria (3):
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Brazil (10):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Panagyurishte
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- China (19):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- Czechia (4):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Ostrava - Vitkovice
  - Research Site, Prague
- France (6):
  - Research Site, Avignon
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, La Tronche
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
- Germany (8):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Gauting
  - Research Site, Gera
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Mainz
  - Research Site, Regensburg
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Székesfehérvár
- Israel (4):
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (6):
  - Research Site, Bergamo
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Roma
  - Research Site, Terni
- Japan (17):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Himeji-shi
  - Research Site, Iwakuni-shi
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Sakaishi
  - Research Site, Sayama
  - Research Site, Tokushima
  - Research Site, Ube-shi
  - Research Site, Yokohama
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Groningen
  - Research Site, Hengelo
  - Research Site, Maastricht
  - Research Site, Rotterdam
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Warsaw
- Romania (3):
  - Research Site, Cluj-Napoca
  - Research Site, Floreşti
  - Research Site, Suceava
- Russia (5):
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Ufa
- Slovakia (6):
  - Research Site, Banská Bystrica
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Nové Zámky
  - Research Site, Trnava
- South Korea (7):
  - Research Site, Changwon
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Badajoz
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Santander
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (10):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kirovohrad
  - Research Site, Kryvyi Rih
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ozguroglu M, Goldman JW, Chen Y, Garassino MC, Medic N, Mann H, Chugh P, Dalvi T, Paz-Ares L. Adverse events self-reported by patients with extensive-stage small-cell lung cancer in the phase III CASPIAN study. Future Oncol. 2025 May;21(12):1511-1523. doi: 10.1080/14796694.2025.2491297. Epub 2025 May 7. PMID 40331625
- [Derived] Xie M, Vuko M, Rodriguez-Canales J, Zimmermann J, Schick M, O'Brien C, Paz-Ares L, Goldman JW, Garassino MC, Gay CM, Heymach JV, Jiang H, Barrett JC, Stewart RA, Lai Z, Byers LA, Rudin CM, Shrestha Y. Molecular classification and biomarkers of outcome with immunotherapy in extensive-stage small-cell lung cancer: analyses of the CASPIAN phase 3 study. Mol Cancer. 2024 May 30;23(1):115. doi: 10.1186/s12943-024-02014-x. PMID 38811992
- [Derived] Goldman JW, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Garassino MC, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Thiyagarajah P, Jiang H, Paz-Ares L; CASPIAN investigators. Durvalumab, with or without tremelimumab, plus platinum-etoposide versus platinum-etoposide alone in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): updated results from a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):51-65. doi: 10.1016/S1470-2045(20)30539-8. Epub 2020 Dec 4. PMID 33285097
- [Derived] Paz-Ares L, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Shire N, Jiang H, Goldman JW; CASPIAN investigators. Durvalumab plus platinum-etoposide versus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): a randomised, controlled, open-label, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1929-1939. doi: 10.1016/S0140-6736(19)32222-6. Epub 2019 Oct 4. PMID 31590988
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00001&attachmentIdentifier=042de696-9399-4abc-8643-673f1237463a&fileName=d419qc00001-csp-v5_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00001&attachmentIdentifier=dafb894c-0f08-4319-a2fe-7389ae3ba87f&fileName=D419qc00001_SAP_Redacted.pdf&versionIdentifier=
- See also: CSPv5_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00001&attachmentIdentifier=11d0f58c-9d10-4c9a-95c3-000528295c1c&fileName=d419qc00001-csp-v5_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in 209 study centers across 23 countries. It included a global cohort (805 patients) and China cohort (188 patients). China cohort comprised 6 patients also in the global cohort and a further 182 patients randomized after end of global cohort recruitment. Results of the global and China cohorts were reported separately.
Pre-assignment Details: Patients were randomized in a 1:1:1 ratio to receive treatment with durvalumab + tremelimumab + etoposide and platinum-based chemotherapy (EP), durvalumab + EP or EP alone. 987 participants were randomized in the study overall. Patients included in both cohorts for Started, Completed and Reasons for Not Completed are not double-counted for participant flow.
Groups:
- All Patients: D + T + EP: During Chemotherapy:
  Patients received durvalumab (D) 1500 milligrams (mg) in combination with tremelimumab (T) 75 mg intravenous (IV) infusion every 3 weeks (Q3W) for 4 doses/cycles (Weeks 0, 3, 6 and 9). For chemotherapy (EP), patients received etoposide (80-100 mg/meters squared [m^2]) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  Post-Chemotherapy:
  Patients then continued to receive durvalumab 1500 mg IV infusion every 4 weeks (Q4W) from Week 12 until progressive disease (PD), unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met. Patients also received an additional dose of tremelimumab 75 mg IV infusion post-chemotherapy (in combination with durvalumab) at Week 16 if they completed all 4 doses of durvalumab + tremelimumab during chemotherapy.
- All Patients: D + EP: During Chemotherapy:
  Patients received durvalumab (D) 1500 mg IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  Post-Chemotherapy:
  Patients then continued to receive durvalumab 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- All Patients: EP: For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). An additional 2 doses of EP (at Weeks 12 and 15) could be given at the investigators' discretion if clinically indicated.
Period: Overall Study
Arm/Group | All Patients: D + T + EP | All Patients: D + EP | All Patients: EP
Started (Randomized in overall study) | 329 | 328 | 330
Randomized and Included in Global Cohort Analysis | 268 | 268 | 269
Received Treatment in Global Cohort | 266 | 265 | 266
Randomized and Included in China Cohort Analysis | 65 | 61 | 62
Received Treatment in China Cohort | 65 | 61 | 62
Included in Both Cohorts (Global + China) | 4 | 1 | 1
Ongoing Study at Global Cohort Final Analysis Data Cut-off (DCO) | 56 | 56 | 31
Ongoing Study at China Cohort Second (Final) Analysis DCO | 16 | 11 | 7
Completed (Ongoing in overall study at long-term follow-up (LTFU) analysis DCO) | 51 | 52 | 18
Not Completed | 278 | 276 | 312
Not completed — Withdrawal by Subject | 6 | 6 | 15
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Death | 270 | 269 | 296

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on the global full analysis set (FAS) (all patients randomized prior to the end of global recruitment) plus the China FAS (all randomized patients in the China cohort). Patients included in both cohorts are not double-counted for the baseline analysis represented by 'All Patients'.
Groups:
- All Patients: D + T + EP: During Chemotherapy:
  Patients received durvalumab (D) 1500 mg in combination with tremelimumab (T) 75 mg IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  Post-Chemotherapy:
  Patients then continued to receive durvalumab 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met. Patients also received an additional dose of tremelimumab 75 mg IV infusion post-chemotherapy (in combination with durvalumab) at Week 16 if they completed all 4 doses of durvalumab + tremelimumab during chemotherapy.
- Total: Total of all reporting groups
Arm/Group | All Patients: D + T + EP | All Patients: D + EP | All Patients: EP | Total
Number analyzed (Participants) | 329 | 328 | 330 | 987
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline data is presented for all patients, as well as separately for the global and China cohorts.
  Participants
    Al Patients: <50 | 21 | 13 | 28 | 62
    Al Patients: ≥50 to <65 | 175 | 195 | 169 | 539
    Al Patients: ≥65 to <75 | 108 | 98 | 110 | 316
    Al Patients: ≥75 | 25 | 22 | 23 | 70
    Global Cohort: number analyzed (Participants) | 268 | 268 | 269 | 805
    Global Cohort: <50 | 16 | 10 | 20 | 46
    Global Cohort: ≥50 to <65 | 138 | 157 | 137 | 432
    Global Cohort: ≥65 to <75 | 91 | 82 | 90 | 263
    Global Cohort: ≥75 | 23 | 19 | 22 | 64
    China Cohort: number analyzed (Participants) | 65 | 61 | 62 | 188
    China Cohort: <50 | 5 | 3 | 8 | 16
    China Cohort: ≥50 to <65 | 40 | 39 | 33 | 112
    China Cohort: ≥65 to <75 | 17 | 16 | 20 | 53
    China Cohort: ≥75 | 3 | 3 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline data is presented for all patients, as well as separately for the global and China cohorts.
  Participants
    All Patients: Female | 74 | 86 | 95 | 255
    All Patients: Male | 255 | 242 | 235 | 732
    Global Cohort: number analyzed (Participants) | 268 | 268 | 269 | 805
    Global Cohort: Female | 66 | 78 | 85 | 229
    Global Cohort: Male | 202 | 190 | 184 | 576
    China Cohort: number analyzed (Participants) | 65 | 61 | 62 | 188
    China Cohort: Female | 8 | 9 | 10 | 27
    China Cohort: Male | 57 | 52 | 52 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline data is presented for all patients, as well as separately for the global and China cohorts.
  Participants
    All Patients: Hispanic or Latino | 7 | 10 | 6 | 23
    All Patients: Not Hispanic or Latino | 321 | 315 | 322 | 958
    All Patients: Unknown or Not Reported | 1 | 3 | 2 | 6
    Global Cohort: number analyzed (Participants) | 268 | 268 | 269 | 805
    Global Cohort: Hispanic or Latino | 7 | 10 | 6 | 23
    Global Cohort: Not Hispanic or Latino | 260 | 255 | 261 | 776
    Global Cohort: Unknown or Not Reported | 1 | 3 | 2 | 6
    China Cohort: number analyzed (Participants) | 65 | 61 | 62 | 188
    China Cohort: Hispanic or Latino | 0 | 0 | 0 | 0
    China Cohort: Not Hispanic or Latino | 65 | 61 | 62 | 188
    China Cohort: Unknown or Not Reported | 0 | 0 | 0 | 0
Race [Count of Participants; unit: Participants] — Population: Baseline data is presented for all patients, as well as separately for the global and China cohorts.
  Participants
    All Patients: White | 215 | 229 | 221 | 665
    All Patients: Black or African American | 1 | 2 | 3 | 6
    All Patients: Asian | 108 | 96 | 103 | 307
    All Patients: Other | 5 | 1 | 2 | 8
    All Patients: Missing | 0 | 0 | 1 | 1
    Global Cohort: number analyzed (Participants) | 268 | 268 | 269 | 805
    Global Cohort: White | 215 | 229 | 221 | 665
    Global Cohort: Black or African American | 1 | 2 | 3 | 6
    Global Cohort: Asian | 47 | 36 | 42 | 125
    Global Cohort: Other | 5 | 1 | 2 | 8
    Global Cohort: Missing | 0 | 0 | 1 | 1
    China Cohort: number analyzed (Participants) | 65 | 61 | 62 | 188
    China Cohort: White | 0 | 0 | 0 | 0
    China Cohort: Black or African American | 0 | 0 | 0 | 0
    China Cohort: Asian | 65 | 61 | 62 | 188
    China Cohort: Other | 0 | 0 | 0 | 0
    China Cohort: Missing | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the Global Cohort; Assessed at Global Cohort Interim Analysis; D + EP Compared With EP
Description: OS was defined as the time from date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. An interim analysis of OS in the global cohort was pre-specified after approximately 318 OS events occurred each between the D + EP and EP groups (60% maturity), and between the D + T + EP and EP groups (60% maturity). At the global cohort interim analysis DCO (11 March 2019), comparison of OS in the D + EP versus (vs) EP groups had crossed the pre-specified boundary. Since these results were considered final in terms of formal statistical testing, they are presented here as a primary outcome measure. Analysis of OS for D + EP vs EP and for D + T + EP vs EP at the time of the global cohort final analysis is presented separately in the subsequent primary outcome measure.
Time Frame: From baseline until death due to any cause. Assessed until global cohort interim analysis DCO (maximum of approximately 23 months).
Population: The global FAS included all patients randomized prior to the end of global recruitment. Interim analysis for OS in the global cohort was performed for comparison of the D + EP vs EP groups only.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Global Cohort: D + EP: During Chemotherapy:
  Patients received durvalumab (D) 1500 mg IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  Post-Chemotherapy:
  Patients then continued to receive durvalumab 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Global Cohort: EP: For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). An additional 2 doses of EP (at Weeks 12 and 15) could be given at the investigators' discretion if clinically indicated.
Arm/Group | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 268 | 269
months | 13.0 [11.5 to 14.8] | 10.3 [9.3 to 11.2]
Statistical Analysis 1: Comparison: Global Cohort: D + EP vs Global Cohort: EP; D + EP vs EP. The global cohort interim analysis of OS was based on a Lan-DeMets alpha spending function with O'Brien Fleming type boundary, using the actual number of events observed as a proportion of the planned total. Boundary for declaring statistical significance was 0.0178 for a 4% overall alpha. Hazard Ratio (HR) <1 favors D + EP to be associated with a longer OS than EP; Test type: Superiority; p = 0.0047, Log Rank — Analysis was performed using the stratified log-rank test, adjusting for planned platinum therapy in Cycle 1 (carboplatin or cisplatin), and using the rank tests of association approach; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.591 to 0.909] — The HR and confidence intervals (CIs) were calculated using a stratified Cox proportional hazards model, adjusting for planned platinum therapy in Cycle 1 (carboplatin or cisplatin), and ties handled by Efron approach

2. Primary Outcome: OS in the Global Cohort; Assessed at Global Cohort Final Analysis; D + EP Compared With EP and D + T + EP Compared With EP
Description: OS was defined as the time from date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. This primary outcome measure presents OS for the analysis of D + EP vs EP and D + T + EP vs EP at the time of the global cohort final analysis DCO (27 January 2020). Analysis of D + EP vs EP at the global cohort interim analysis DCO is presented in the previous primary outcome measure. Analysis of D + T + EP vs D + EP (global cohort final analysis) is presented as a secondary outcome measure.
Time Frame: From baseline until death due to any cause. Assessed until global cohort final analysis DCO (maximum of approximately 33 months).
Population: The global FAS included all patients randomized prior to the end of global recruitment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Global Cohort: D + T + EP: During Chemotherapy:
  Patients received durvalumab (D) 1500 mg in combination with tremelimumab (T) 75 mg IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  Post-Chemotherapy:
  Patients then continued to receive durvalumab 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met. Patients also received an additional dose of tremelimumab 75 mg IV infusion post-chemotherapy (in combination with durvalumab) at Week 16 if they completed all 4 doses of durvalumab + tremelimumab during chemotherapy.
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 268 | 268 | 269
months | 10.4 [9.6 to 12.0] | 12.9 [11.3 to 14.7] | 10.5 [9.3 to 11.2]
Statistical Analysis 1: Comparison: Global Cohort: D + EP vs Global Cohort: EP; D + EP vs EP. HR <1 favors D + EP to be associated with a longer OS than EP; Test type: Superiority; p = 0.0032, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.625 to 0.910] — The HR and CIs were calculated using a stratified Cox proportional hazards model, adjusting for planned platinum therapy in Cycle 1 (carboplatin or cisplatin), and ties handled by Efron approach
Statistical Analysis 2: Comparison: Global Cohort: D + T + EP vs Global Cohort: EP; D + T + EP vs EP. The alpha level applied at the global cohort final analysis was adjusted (using a generalized Haybittle-Peto method) to account for actual alpha spent at the interim analysis based on the actual final total number of events, and thus maintain control of overall Type I error. Boundary for declaring statistical significance was 0.0418 for a 5% overall alpha. HR <1 favors D + T + EP to be associated with a longer OS than EP; Test type: Superiority; p = 0.0451, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.682 to 0.995] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: OS in the China Cohort; Assessed at China Cohort First Analysis; D + EP Compared With EP
Description: OS was defined as the time from date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. An analysis of OS for D + EP vs EP in the China cohort was pre-specified at approximately 60% maturity (to ensure a similar maturity to the interim analysis of the Global cohort). This primary outcome measure presents OS for analysis of D + EP vs EP at the China cohort first analysis DCO (06 January 2020), and is comparable in terms of maturity with the interim analysis of OS for D + EP vs EP in the Global cohort. Analysis of OS for D + EP vs EP and for D + T + EP vs EP at the time of the China cohort second analysis is presented separately in the subsequent primary outcome measure.
Time Frame: From baseline until death due to any cause. Assessed until China cohort first analysis DCO (maximum of approximately 19 months).
Population: The China FAS included all randomized patients in the China cohort. China cohort first analysis for OS was performed for comparison of the D + EP vs EP groups only.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- China Cohort: D + EP: During Chemotherapy:
  Patients received durvalumab (D) 1500 mg IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  Post-Chemotherapy:
  Patients then continued to receive durvalumab 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- China Cohort: EP: For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). An additional 2 doses of EP (at Weeks 12 and 15) could be given at the investigators' discretion if clinically indicated.
Arm/Group | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 61 | 62
months | 14.4 [12.3 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 10.9 [8.9 to 14.0]
Statistical Analysis 1: Comparison: China Cohort: D + EP vs China Cohort: EP; D + EP vs EP. HR <1 favors D + EP to be associated with a longer OS than EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.0664, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.414 to 1.029] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: OS in the China Cohort; Assessed at China Cohort Second Analysis; D + EP Compared With EP and D + T + EP Compared With EP
Description: OS was defined as the time from date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. An analysis of OS for D + T + EP vs EP in the China cohort was pre-specified at approximately 80% maturity (to ensure a similar maturity to the final analysis of the Global cohort). This primary outcome measure presents OS for analysis of D + EP vs EP and D + T + EP vs EP at the time of the China cohort second analysis DCO (02 November 2020), and is comparable in terms of maturity with the final analysis of OS for D + EP vs EP and D + T + EP vs EP in the Global cohort. Analysis of D + EP vs EP at the China cohort first analysis DCO is presented in the previous primary outcome measure. Analysis of D + T + EP vs D + EP (China cohort second analysis) is presented as a secondary outcome measure.
Time Frame: From baseline until death due to any cause. Assessed until China cohort second analysis DCO (maximum of approximately 29 months).
Population: The China FAS included all randomized patients in the China cohort.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- China Cohort: D + T + EP: During Chemotherapy:
  Patients received durvalumab (D) 1500 mg in combination with tremelimumab (T) 75 mg IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). For chemotherapy (EP), patients received etoposide (80-100 mg/m^2) with either carboplatin (area under the curve 5-6) or cisplatin (75-80 mg/m^2) IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  Post-Chemotherapy:
  Patients then continued to receive durvalumab 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met. Patients also received an additional dose of tremelimumab 75 mg IV infusion post-chemotherapy (in combination with durvalumab) at Week 16 if they completed all 4 doses of durvalumab + tremelimumab during chemotherapy.
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
months | 16.1 [11.3 to 18.6] | 14.4 [12.3 to 17.0] | 10.9 [8.9 to 14.0]
Statistical Analysis 1: Comparison: China Cohort: D + EP vs China Cohort: EP; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.1455, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.504 to 1.106] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: China Cohort: D + T + EP vs China Cohort: EP; D + T + EP vs EP. HR <1 favors D + T + EP to be associated with a longer OS than EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.0314, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.439 to 0.964] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: OS in the Global Cohort; D + T + EP Compared With D + EP
Description: OS was defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. This secondary outcome measure presents OS for the analysis of D + T + EP vs D + EP in the global cohort. The alternative treatment comparisons in the global cohort were performed as primary outcome measures.
Time Frame: as for outcome 2
Population: The global FAS included all patients randomized prior to the end of global recruitment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP
Number analyzed (Participants) | 268 | 268
months | 10.4 [9.6 to 12.0] | 12.9 [11.3 to 14.7]
Statistical Analysis 1: Comparison: Global Cohort: D + T + EP vs Global Cohort: D + EP; D + T + EP vs D + EP. HR <1 favors D + T + EP to be associated with a longer OS than D + EP; Test type: Superiority; p = 0.4352, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.890 to 1.309] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Progression-Free Survival (PFS) in the Global Cohort
Description: PFS (per Response Evaluation Criteria in Solid Tumors, version 1.1 [RECIST 1.1] using Investigator assessments) was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression. Progression (ie, PD) was defined as at least a 20% increase in the sum of diameters of target lesions (TLs), taking as reference the smallest previous sum of diameters (nadir) and an absolute increase of ≥5 millimeters (mm) for the sum from nadir. For evaluation of non-target lesions (NTLs), PD was defined as unequivocal progression of existing NTLs. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline, Week 6, Week 12 then every 8 weeks relative to the date of randomization until RECIST 1.1-defined progression. Assessed until global cohort final analysis DCO (maximum of approximately 33 months).
Population: The global FAS included all patients randomized prior to the end of global recruitment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 268 | 268 | 269
months | 4.9 [4.7 to 5.9] | 5.1 [4.7 to 6.2] | 5.4 [4.8 to 6.2]
Statistical Analysis 1: Comparison: Global Cohort: D + EP vs Global Cohort: EP; D + EP vs EP. HR <1 favors D + EP to be associated with a longer PFS than EP; Test type: Superiority; p = 0.0157, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.665 to 0.959] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Global Cohort: D + T + EP vs Global Cohort: EP; D + T + EP vs EP. HR <1 favors D + T + EP to be associated with a longer PFS than EP; Test type: Superiority; p = 0.0568, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.696 to 1.005] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Global Cohort: D + T + EP vs Global Cohort: D + EP; D + T + EP vs D + EP. HR <1 favors D + T + EP to be associated with a longer PFS than D + EP; Test type: Superiority; p = 0.7540, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.857 to 1.235] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Objective Response Rate (ORR) in the Global Cohort
Description: ORR (per RECIST 1.1 using Investigator assessments) was defined as the percentage of patients with at least 1 visit response of Complete Response (CR) or Partial Response (PR). CR was defined as disappearance of all TLs since baseline (any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm) or disappearance of all NTLs since baseline (all lymph nodes must be non-pathological in size [<10 mm short axis]). PR was defined as at least a 30% decrease in the sum of diameters of TLs (taking as reference the baseline sum of diameters).
Time Frame: as for outcome 6
Population: The global FAS included all patients randomized prior to the end of global recruitment. The denominator was a subset of the FAS population who had measurable disease at baseline.
Measure: Number; unit: percentage of patients
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 267 | 268 | 269
percentage of patients | 74.2 | 79.5 | 70.6
Statistical Analysis 1: Comparison: Global Cohort: D + EP vs Global Cohort: EP; D + EP vs EP. An odds ratio >1 favors D + EP; Test type: Superiority; p = 0.0177, Regression, Logistic — Analysis was performed using a logistic regression model, adjusting for planned platinum therapy in Cycle 1 (carboplatin or cisplatin). P-value is based on twice the change in log-likelihood resulting from addition of a treatment factor to the model; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.086 to 2.401]
Statistical Analysis 2: Comparison: Global Cohort: D + T + EP vs Global Cohort: EP; D + T + EP vs EP. An odds ratio >1 favors D + T + EP; Test type: Superiority; p = 0.3611, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.817 to 1.746]

8. Secondary Outcome: Percentage of Patients Alive and Progression Free at 6 Months (APF6) in the Global Cohort
Description: The APF6 was defined as the percentage of patients who were alive and progression free at 6 months from randomization (ie, PFS rate at 6 months). PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline, Week 6, Week 12 then every 8 weeks relative to the date of randomization until RECIST 1.1-defined progression. Assessed until 6 months post-randomization.
Population: The global FAS included all patients randomized prior to the end of global recruitment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 268 | 268 | 269
percentage of patients | 43.2 [37.1 to 49.1] | 45.4 [39.3 to 51.3] | 45.8 [39.5 to 51.9]

9. Secondary Outcome: Percentage of Patients Alive and Progression Free at 12 Months (APF12) in the Global Cohort
Description: The APF12 was defined as the percentage of patients who were alive and progression free at 12 months from randomization (ie, PFS rate at 12 months). PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline, Week 6, Week 12 then every 8 weeks relative to the date of randomization until RECIST 1.1-defined progression. Assessed until 12 months post-randomization.
Population: The global FAS included all patients randomized prior to the end of global recruitment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 268 | 268 | 269
percentage of patients | 16.9 [12.6 to 21.7] | 17.9 [13.5 to 22.8] | 5.3 [2.9 to 8.8]

10. Secondary Outcome: Percentage of Patients Alive at 18 Months (OS18) in the Global Cohort
Description: OS18 was defined as the percentage of patients who were alive at 18 months after randomization per the Kaplan-Meier estimate of OS at 18 months.
Time Frame: At 18 months post-randomization. Assessed at the global cohort final analysis DCO (27 January 2020).
Population: The global FAS included all patients randomized prior to the end of global recruitment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 268 | 268 | 269
percentage of patients | 30.7 [25.2 to 36.4] | 32.0 [26.5 to 37.7] | 24.8 [19.7 to 30.1]

11. Secondary Outcome: Pharmacokinetics (PK) of Durvalumab; Peak and Trough Serum Concentrations in the Global Cohort
Description: To evaluate PK, blood samples were collected at pre-specified timepoints and peak and trough serum concentrations of durvalumab were determined. Peak concentration on Week 0 is the post-infusion concentration of Week 0 (collected within 10 minutes of the end of infusion). Trough concentrations on Weeks 3 and 12 are the pre-infusion concentrations of Weeks 3 and 12, respectively.
Time Frame: Samples were collected post-dose on Day 1 (Week 0), and pre-dose on Weeks 3 and 12. Assessed at the global cohort final analysis DCO (27 January 2020).
Population: The global PK analysis set included all patients randomized prior to the end of global recruitment who received at least 1 dose of investigational product (IP), per the protocol for whom any post-dose PK data were available. PK for durvalumab was performed for the D + T + EP and D + EP groups only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (μg/mL)
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP
Number analyzed (Participants) | 257 | 261
micrograms/milliliter (μg/mL)
  Week 0: peak concentration: number analyzed (Participants) | 239 | 226
  Week 0: peak concentration | 447.3 (78.21) | 502.6 (30.52)
  Week 3: trough concentration: number analyzed (Participants) | 232 | 237
  Week 3: trough concentration | 91.86 (74.36) | 109.5 (64.55)
  Week 12: trough concentration: number analyzed (Participants) | 173 | 200
  Week 12: trough concentration | 199.2 (49.58) | 239.3 (50.68)

12. Secondary Outcome: PK of Tremelimumab; Peak and Trough Serum Concentrations in the Global Cohort
Description: To evaluate PK, blood samples were collected at pre-specified timepoints and peak and trough serum concentrations of tremelimumab were determined. Peak concentration on Week 0 is the post-infusion concentration of Week 0 (collected within 10 minutes of the end of infusion). Trough concentrations on Weeks 3 and 12 are the pre-infusion concentrations of Weeks 3 and 12, respectively.
Time Frame: as for outcome 11
Population: The global PK analysis set included all patients randomized prior to the end of global recruitment who received at least 1 dose of IP, per the protocol for whom any post-dose PK data were available. PK for tremelimumab was performed for the D + T + EP group only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Global Cohort: D + T + EP
Number analyzed (Participants) | 257
μg/mL
  Week 0: peak concentration: number analyzed (Participants) | 236
  Week 0: peak concentration | 22.77 (52.15)
  Week 3: trough concentration: number analyzed (Participants) | 227
  Week 3: trough concentration | 4.245 (81.68)
  Week 12: trough concentration: number analyzed (Participants) | 148
  Week 12: trough concentration | 7.576 (59.25)

13. Secondary Outcome: Number of Patients With Anti-Drug Antibody (ADA) Response to Durvalumab in the Global Cohort
Description: Serum sampling for ADA assessment was conducted utilizing a tiered approach (screen, confirm, titer). ADA positive post-baseline only was also referred to as treatment-induced ADA. Treatment-emergent ADA was defined as the sum of treatment-induced ADA and treatment-boosted ADA (defined as baseline positive ADA titer that was boosted to ≥4-fold during the study period). Persistently positive was defined as having ≥2 post-baseline ADA positive measurements with ≥16 weeks between first and last positive, or an ADA positive result at the last available assessment. Transiently positive was defined as having ≥1 post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. Presence of neutralizing antibody (nAb) was tested for all ADA positive samples. Results are reported as number of patients with ADA responses to durvalumab for each indicated category.
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of IP (ie, durvalumab). Assessed at the global cohort final analysis DCO (27 January 2020).
Population: The global ADA evaluable patients included those in the global safety analysis set who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result. ADA for durvalumab was performed for the D + T + EP and D + EP groups only. The denominator was durvalumab ADA evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP
Number analyzed (Participants) | 191 | 205
Participants
  ADA positive at any visit (ADA prevalence) | 6 | 11
  Treatment-emergent ADA positive (ADA incidence) | 0 | 0
  Treatment-boosted ADA | 0 | 0
  Treatment-induced ADA (ADA positive post-baseline only) | 0 | 0
  ADA positive at baseline only | 6 | 11
  ADA positive post-baseline and positive at baseline | 0 | 0
  Persistently positive | 0 | 0
  Transiently positive | 0 | 0
  nAb positive at any visit | 1 | 0

14. Secondary Outcome: Number of Patients With ADA Response to Tremelimumab in the Global Cohort
Description: Serum sampling for ADA assessment was conducted utilizing a tiered approach (screen, confirm, titer). ADA positive post-baseline only was also referred to as treatment-induced ADA. Treatment-emergent ADA (or ADA incidence) was defined as the sum of treatment-induced ADA and treatment-boosted ADA (defined as baseline positive ADA titer that was boosted to ≥4-fold during the study period). Persistently positive was defined as having ≥2 post-baseline ADA positive measurements with ≥16 weeks between first and last positive, or an ADA positive result at the last available assessment. Transiently positive was defined as having ≥1 post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. The presence of nAb was tested for all ADA positive samples. Results are reported as number of patients with ADA responses to tremelimumab for each indicated category.
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of IP (ie, tremelimumab). Assessed at the global cohort final analysis DCO (27 January 2020).
Population: The global ADA evaluable patients included those in the global safety analysis set who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result. ADA for tremelimumab was performed for the D + T + EP group only. The denominator was tremelimumab ADA evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Global Cohort: D + T + EP
Number analyzed (Participants) | 178
Participants
  ADA positive at any visit (ADA prevalence) | 11
  Treatment-emergent ADA positive (ADA incidence) | 5
  Treatment-boosted ADA | 0
  Treatment-induced ADA (ADA positive post-baseline only) | 5
  ADA positive at baseline only | 6
  ADA positive post-baseline and positive at baseline | 0
  Persistently positive | 4
  Transiently positive | 1
  nAb positive at any visit | 2

15. Secondary Outcome: Time to Deterioration of Health-Related Quality of Life (HRQoL) and Patient Reported Outcome (PRO) Symptoms, Assessed Using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) in the Global Cohort
Description: The EORTC QLQ-Core 30 version 3 (QLQ-C30 v3) was included for assessing HRQoL. It assesses HRQoL/health status through 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), and a global health and QoL scale. 6 single-item symptom measures are also included: dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. Scores from 0 to 100 were derived for each of the 15 domains, with higher scores representing greater functioning, greater HRQoL, or greater level of symptoms. Time to deterioration (calculated using the Kaplan-Meier technique) was defined as time from randomization until the date of first clinically meaningful deterioration (a decrease in score from baseline of ≥10) that is confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration.
Time Frame: At baseline, Weeks 3, 6, 9, 12, 16 and 20, then Q4W until PD, on Day 28 and 2 months post-PD, then every 8 weeks until second progression/death (whichever comes first). Assessed until global cohort final analysis DCO (maximum of approximately 33 months).
Population: The global FAS included all patients randomized prior to the end of global recruitment. For QLQ-C30 function scales and global health status/HRQoL, only patients with baseline scores ≥10 (and with data available) were included in the analysis. For QLQ-C30 symptom scales/items, only patients with baseline scores ≤90 (and with data available) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 262 | 261 | 260
months
  QLQ-C30 Global Health Status / HRQoL: number analyzed (Participants) | 247 | 239 | 232
  QLQ-C30 Global Health Status / HRQoL | 7.2 [5.8 to 8.3] | 8.4 [7.3 to 11.0] | 7.4 [6.5 to 9.3]
  QLQ-C30 Cognitive Functioning: number analyzed (Participants) | 251 | 245 | 242
  QLQ-C30 Cognitive Functioning | 6.0 [5.0 to 7.0] | 8.4 [7.3 to 10.3] | 6.0 [5.2 to 7.1]
  QLQ-C30 Emotional Functioning: number analyzed (Participants) | 248 | 242 | 240
  QLQ-C30 Emotional Functioning | 7.6 [6.6 to 9.5] | 11.8 [8.6 to 16.6] | 7.3 [6.7 to 8.3]
  QLQ-C30 Physical Functioning: number analyzed (Participants) | 247 | 244 | 240
  QLQ-C30 Physical Functioning | 6.0 [5.0 to 6.9] | 8.4 [7.4 to 12.0] | 6.5 [6.0 to 8.2]
  QLQ-C30 Role Functioning: number analyzed (Participants) | 236 | 231 | 226
  QLQ-C30 Role Functioning | 5.0 [4.1 to 6.5] | 7.4 [5.7 to 10.2] | 5.9 [4.5 to 6.7]
  QLQ-C30 Social Functioning: number analyzed (Participants) | 244 | 237 | 236
  QLQ-C30 Social Functioning | 6.2 [5.0 to 7.4] | 7.4 [6.5 to 8.8] | 6.3 [4.9 to 7.4]
  QLQ-C30 Fatigue: number analyzed (Participants) | 242 | 244 | 232
  QLQ-C30 Fatigue | 4.2 [3.1 to 4.7] | 5.5 [4.0 to 6.6] | 4.5 [3.5 to 5.3]
  QLQ-C30 Nausea / Vomiting: number analyzed (Participants) | 252 | 245 | 244
  QLQ-C30 Nausea / Vomiting | 7.5 [6.1 to 8.6] | 8.4 [6.6 to 10.2] | 6.6 [5.6 to 7.5]
  QLQ-C30 Pain: number analyzed (Participants) | 243 | 240 | 233
  QLQ-C30 Pain | 6.9 [6.0 to 7.7] | 8.0 [6.8 to 10.4] | 6.7 [6.2 to 7.8]
  QLQ-C30 Appetite Loss: number analyzed (Participants) | 236 | 231 | 224
  QLQ-C30 Appetite Loss | 6.9 [5.6 to 8.5] | 8.3 [6.8 to 11.0] | 6.6 [5.5 to 7.5]
  QLQ-C30 Constipation: number analyzed (Participants) | 243 | 240 | 229
  QLQ-C30 Constipation | 8.5 [7.1 to 10.8] | 11.5 [8.3 to 14.7] | 7.3 [6.2 to 9.0]
  QLQ-C30 Diarrhea: number analyzed (Participants) | 250 | 244 | 244
  QLQ-C30 Diarrhea | 8.9 [7.5 to 10.8] | 14.7 [9.4 to 21.1] | 7.7 [7.1 to 9.5]
  QLQ-C30 Dyspnea: number analyzed (Participants) | 227 | 225 | 218
  QLQ-C30 Dyspnea | 7.2 [5.6 to 8.3] | 9.0 [7.6 to 12.7] | 7.5 [6.6 to 9.0]
  QLQ-C30 Insomnia: number analyzed (Participants) | 226 | 226 | 210
  QLQ-C30 Insomnia | 7.1 [6.1 to 8.6] | 8.6 [7.1 to 11.8] | 7.3 [6.4 to 8.3]

16. Secondary Outcome: Time to Deterioration of PRO Symptoms, Assessed Using EORTC QLQ-Lung Cancer Module 13 (QLQ-LC13) in the Global Cohort
Description: The EORTC QLQ-LC13 is a disease-specific 13-item self-administered questionnaire for lung cancer, to be used in conjunction with the EORTC QLQ-C30. It comprises both multi-item and single-item measures of lung cancer-associated symptoms (ie, coughing, hemoptysis, dyspnea, and pain) and side effects from conventional chemotherapy and radiotherapy (ie, hair loss, neuropathy, sore mouth, and dysphagia). Scores from 0 to 100 were derived for each symptom item, with higher scores representing greater level of symptoms. Time to deterioration (calculated using the Kaplan-Meier technique) was defined as time from randomization until the date of first clinically meaningful deterioration (an increase in score from baseline of ≥10) that is confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration.
Time Frame: as for outcome 15
Population: The global FAS included all patients randomized prior to the end of global recruitment. For QLQ-L13 symptom scales/items, only patients with baseline scores ≤90 (and with data available) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 262 | 261 | 260
months
  QLQ-LC13 Coughing: number analyzed (Participants) | 233 | 230 | 230
  QLQ-LC13 Coughing | 7.7 [6.9 to 10.8] | 9.3 [8.0 to 14.1] | 7.7 [6.7 to 9.5]
  QLQ-LC13 Dyspnea: number analyzed (Participants) | 249 | 241 | 240
  QLQ-LC13 Dyspnea | 6.3 [4.9 to 7.4] | 6.5 [5.5 to 7.8] | 5.5 [4.6 to 7.2]
  QLQ-LC13 Hemoptysis: number analyzed (Participants) | 252 | 243 | 245
  QLQ-LC13 Hemoptysis | 11.4 [8.9 to 18.6] | 18.3 [14.5 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 10.8 [8.4 to 11.9]
  QLQ-LC13 Pain in Arm or Shoulder: number analyzed (Participants) | 245 | 241 | 238
  QLQ-LC13 Pain in Arm or Shoulder | 7.1 [6.3 to 8.3] | 9.7 [8.1 to 15.1] | 7.6 [6.6 to 9.3]
  QLQ-LC13 Pain in Chest: number analyzed (Participants) | 243 | 239 | 240
  QLQ-LC13 Pain in Chest | 8.5 [7.2 to 10.8] | 11.5 [8.4 to 15.8] | 7.9 [7.2 to 9.9]
  QLQ-LC13 Pain in Other Parts: number analyzed (Participants) | 245 | 236 | 231
  QLQ-LC13 Pain in Other Parts | 7.4 [6.5 to 8.7] | 7.8 [6.6 to 9.3] | 6.6 [5.1 to 7.5]

17. Secondary Outcome: Change From Baseline in Primary PRO Symptoms as Assessed by EORTC QLQ in the Global Cohort; D + T + EP Compared With EP
Description: A mixed model repeated measures (MMRM) analysis of EORTC QLQ-C30 and EORTC QLQ-LC13 was performed for 5 primary PRO symptoms (cough, dyspnea, chest pain, fatigue and appetite loss), and considered all data from baseline to PD or 12 months, excluding visits with excessive missing data (defined as >75% missing data). An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items, with higher scores representing greater symptom severity. An improvement in symptoms was indicated by a negative change from baseline. A positive change from baseline indicated a deterioration of symptoms. A minimum clinically meaningful change was defined as an absolute change from baseline of ≥10. This outcome measure presents change from baseline for primary PRO symptoms (reported as adjusted means) for analysis of D + T + EP vs P. Analysis of D + EP vs EP is presented in a separate outcome measure.
Time Frame: At baseline, Weeks 3, 6, 9, 12, 16 and 20, then Q4W until PD, on Day 28 and 2 months post-PD, then every 8 weeks until second progression/death (whichever comes first). Assessed up to 12 months.
Population: The global FAS included all patients randomized prior to the end of global recruitment. For each symptom scale, only patients with data available were included in the analysis.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Global Cohort: D + T + EP | Global Cohort: EP
Number analyzed (Participants) | 262 | 260
scores on a scale
  EORTC QLQ-LC13 Cough: number analyzed (Participants) | 239 | 232
  EORTC QLQ-LC13 Cough | -15.1 (1.74) | -14.6 (1.76)
  EORTC QLQ-LC13 Dyspnea: number analyzed (Participants) | 239 | 232
  EORTC QLQ-LC13 Dyspnea | -6.8 (1.60) | -6.6 (1.62)
  EORTC QLQ-LC13 Chest pain: number analyzed (Participants) | 239 | 232
  EORTC QLQ-LC13 Chest pain | -7.4 (1.65) | -7.0 (1.67)
  EORTC QLQ-C30 Fatigue: number analyzed (Participants) | 239 | 233
  EORTC QLQ-C30 Fatigue | -6.1 (1.84) | -6.3 (1.86)
  EORTC QLQ-C30 Appetite loss: number analyzed (Participants) | 239 | 233
  EORTC QLQ-C30 Appetite loss | -8.7 (2.02) | -9.5 (2.05)

18. Secondary Outcome: Change From Baseline in Primary Symptoms, Assessed Using EORTC QLQ-C30 and EORTC QLQ-LC13 in the Global Cohort; D + EP Compared With EP
Description: A MMRM analysis of EORTC QLQ-C30 and EORTC QLQ-LC13 was performed for 5 primary PRO symptoms (cough, dyspnea, chest pain, fatigue and appetite loss), and considered all data from baseline to PD or 12 months, excluding visits with excessive missing data (defined as >75% missing data). An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items, with higher scores representing greater symptom severity. An improvement in symptoms was indicated by a negative change from baseline. A positive change from baseline indicated a deterioration of symptoms. A minimum clinically meaningful change was defined as an absolute change from baseline of ≥10. This outcome measure presents change from baseline for primary PRO symptoms (reported as adjusted means) for analysis of D + EP vs EP. Analysis of D + T + EP vs EP is presented in a separate outcome measure.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Global Cohort: D + EP | Global Cohort: EP
Number analyzed (Participants) | 261 | 260
scores on a scale
  EORTC QLQ-LC13 Cough: number analyzed (Participants) | 232 | 232
  EORTC QLQ-LC13 Cough | -15.0 (1.64) | -15.4 (1.72)
  EORTC QLQ-LC13 Dyspnea: number analyzed (Participants) | 232 | 232
  EORTC QLQ-LC13 Dyspnea | -7.1 (1.44) | -6.5 (1.50)
  EORTC QLQ-LC13 Chest pain: number analyzed (Participants) | 232 | 232
  EORTC QLQ-LC13 Chest pain | -7.8 (1.59) | -7.2 (1.65)
  EORTC QLQ-C30 Fatigue: number analyzed (Participants) | 233 | 233
  EORTC QLQ-C30 Fatigue | -5.8 (1.62) | -4.5 (1.69)
  EORTC QLQ-C30 Appetite loss: number analyzed (Participants) | 233 | 233
  EORTC QLQ-C30 Appetite loss | -10.1 (1.73) | -7.6 (1.81)

19. Secondary Outcome: OS in the China Cohort; D + T + EP Compared With D + EP
Description: OS was defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. This secondary outcome measure presents OS for the analysis of D + T + EP vs D + EP at the China cohort second analysis DCO (02 November 2020). The alternative treatment comparisons were performed as primary outcome measures.
Time Frame: as for outcome 4
Population: The China FAS included all randomized patients in the China cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP
Number analyzed (Participants) | 65 | 61
months | 16.1 [11.3 to 18.6] | 14.4 [12.3 to 17.0]
Statistical Analysis 1: Comparison: China Cohort: D + T + EP vs China Cohort: D + EP; D + T + EP vs D + EP. HR <1 favors D + T + EP to be associated with a longer OS than D + EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.4470, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.574 to 1.277] — [estimate comment as in outcome 2, analysis 1]

20. Secondary Outcome: PFS in the China Cohort
Description: PFS (per RECIST 1.1 using Investigator assessments) was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression. Progression (ie, PD) was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir) and an absolute increase of ≥5 mm for the sum from nadir. For evaluation of NTLs, PD was defined as unequivocal progression of existing NTLs. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline, Week 6, Week 12 then every 8 weeks relative to the date of randomization until RECIST 1.1-defined progression. Assessed until China cohort second analysis DCO (maximum of approximately 29 months).
Population: The China FAS included all randomized patients in the China cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
months | 5.6 [4.8 to 6.6] | 4.9 [4.7 to 5.5] | 5.5 [4.9 to 6.3]
Statistical Analysis 1: Comparison: China Cohort: D + EP vs China Cohort: EP; D + EP vs EP. HR <1 favors D + EP to be associated with a longer PFS than EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.8934, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.661 to 1.437] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: China Cohort: D + T + EP vs China Cohort: EP; D + T + EP vs EP. HR <1 favors D + T + EP to be associated with a longer PFS than EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.1035, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.487 to 1.068] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: China Cohort: D + T + EP vs China Cohort: D + EP; D + T + EP vs D + EP. HR <1 favors D + T + EP to be associated with a longer PFS than D + EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.1673, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.522 to 1.116] — [estimate comment as in outcome 2, analysis 1]

21. Secondary Outcome: ORR in the China Cohort
Description: ORR (per RECIST 1.1 using Investigator assessments) was defined as the percentage of patients with at least 1 visit response of CR or PR. CR was defined as disappearance of all TLs since baseline (any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm) or disappearance of all NTLs since baseline (all lymph nodes must be non-pathological in size [<10 mm short axis]). PR was defined as at least a 30% decrease in the sum of diameters of TLs (taking as reference the baseline sum of diameters).
Time Frame: as for outcome 20
Population: The China FAS included all randomized patients in the China cohort.
Measure: Number; unit: percentage of patients
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
percentage of patients | 84.6 | 78.7 | 72.6
Statistical Analysis 1: Comparison: China Cohort: D + EP vs China Cohort: EP; D + EP vs EP. An odds ratio >1 favors D + EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.4320, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.610 to 3.244]
Statistical Analysis 2: Comparison: China Cohort: D + T + EP vs China Cohort: EP; D + T + EP vs EP. An odds ratio >1 favors D + T + EP. The study was not designed or powered to show statistical significance for efficacy endpoints in the China cohort, so all statistical analyses for the China cohort were considered exploratory; Test type: Other; p = 0.0986, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.874 to 5.118]

22. Secondary Outcome: APF6 in the China Cohort
Description: as for outcome 8
Time Frame: as for outcome 8
Population: The China FAS included all randomized patients in the China cohort.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
percentage of patients | 43.7 [31.2 to 55.5] | 35.2 [23.3 to 47.4] | 43.1 [29.8 to 55.7]

23. Secondary Outcome: APF12 in the China Cohort
Description: as for outcome 9
Time Frame: as for outcome 9
Population: The China FAS included all randomized patients in the China cohort.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
percentage of patients | 21.0 [12.0 to 31.9] | 12.3 [5.4 to 22.2] | 6.2 [1.6 to 15.3]

24. Secondary Outcome: OS18 in the China Cohort
Description: as for outcome 10
Time Frame: At 18 months post-randomization. Assessed at the China cohort second analysis DCO (02 November 2020).
Population: The China FAS included all randomized patients in the China cohort.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
percentage of patients | 40.0 [28.1 to 51.6] | 36.1 [24.3 to 48.0] | 23.4 [13.6 to 34.6]

25. Secondary Outcome: PK of Durvalumab; Peak and Trough Serum Concentrations in the China Cohort
Description: as for outcome 11
Time Frame: Samples were collected post-dose on Day 1 (Week 0), and pre-dose on Weeks 3 and 12. Assessed at the China cohort second analysis DCO (02 November 2020).
Population: The China PK analysis set included all patients in the China cohort who received at least 1 dose of IP, per the protocol for whom any post-dose PK data were available. PK for durvalumab was performed for the D + T + EP and D + EP groups only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP
Number analyzed (Participants) | 64 | 59
μg/mL
  Week 0: peak concentration | 429.4 (19.49) | 432.0 (91.79)
  Week 3: trough concentration: number analyzed (Participants) | 61 | 54
  Week 3: trough concentration | 81.21 (46.14) | 96.24 (64.44)
  Week 12: trough concentration: number analyzed (Participants) | 46 | 50
  Week 12: trough concentration | 151.0 (29.82) | 194.4 (53.34)

26. Secondary Outcome: PK of Tremelimumab; Peak and Trough Serum Concentrations in the China Cohort
Description: as for outcome 12
Time Frame: as for outcome 25
Population: The China PK analysis set included all patients in the China cohort who received at least 1 dose of IP, per the protocol for whom any post-dose PK data were available. PK for tremelimumab was performed for the D + T + EP group only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | China Cohort: D + T + EP
Number analyzed (Participants) | 64
μg/mL
  Week 0: peak concentration | 24.34 (27.05)
  Week 3: trough concentration: number analyzed (Participants) | 61
  Week 3: trough concentration | 4.530 (60.60)
  Week 12: trough concentration: number analyzed (Participants) | 45
  Week 12: trough concentration | 9.523 (43.94)

27. Secondary Outcome: Number of Patients With ADA Response to Durvalumab in the China Cohort
Description: Serum sampling for ADA assessment was conducted utilizing a tiered approach (screen, confirm, titer). ADA positive post-baseline only was also referred to as treatment-induced ADA. Treatment-emergent ADA was defined as the sum of treatment-induced ADA and treatment-boosted ADA (defined as baseline positive ADA titer that was boosted to ≥4-fold during the study period). Persistently positive was defined as having ≥2 post-baseline ADA positive measurements with ≥16 weeks between first and last positive, or an ADA positive result at the last available assessment. Transiently positive was defined as having ≥1 post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. Presence of nAb was tested for all ADA positive samples. Results are reported as number of patients with ADA responses to durvalumab for each indicated category.
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of IP (ie, durvalumab). Assessed at the China cohort second analysis DCO (02 November 2020).
Population: The China ADA evaluable patients included those in the China safety analysis set who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result. ADA for durvalumab was performed for the D + T + EP and D + EP groups only. The denominator was durvalumab ADA evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP
Number analyzed (Participants) | 53 | 51
Participants
  ADA positive at any visit (ADA prevalence) | 0 | 0
  Treatment-emergent ADA positive (ADA incidence) | 0 | 0
  Treatment-boosted ADA | 0 | 0
  Treatment-induced ADA (ADA positive post-baseline only) | 0 | 0
  ADA positive at baseline only | 0 | 0
  ADA positive post-baseline and positive at baseline | 0 | 0
  Persistently positive | 0 | 0
  Transiently positive | 0 | 0
  nAb positive at any visit | 0 | 0

28. Secondary Outcome: Number of Patients With ADA Response to Tremelimumab in the China Cohort
Description: as for outcome 14
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of IP (ie, tremelimumab). Assessed at the China cohort second analysis DCO (02 November 2020).
Population: The China ADA evaluable patients included those in the China safety analysis set who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result. ADA for tremelimumab was performed for the D + T + EP group only. The denominator was tremelimumab ADA evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | China Cohort: D + T + EP
Number analyzed (Participants) | 51
Participants
  ADA positive at any visit (ADA prevalence) | 3
  Treatment-emergent ADA positive (ADA incidence) | 3
  Treatment-boosted ADA | 0
  Treatment-induced ADA (ADA positive post-baseline only) | 3
  ADA positive at baseline only | 0
  ADA positive post-baseline and positive at baseline | 0
  Persistently positive | 3
  Transiently positive | 0
  nAb positive at any visit | 0

29. Secondary Outcome: Time to Deterioration of HRQoL and PRO Symptoms, Assessed Using EORTC QLQ in the China Cohort
Description: The EORTC QLQ-C30 v3 was included for assessing HRQoL. It assesses HRQoL/health status through 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), and a global health and QoL scale. 6 single-item symptom measures are also included: dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. Scores from 0 to 100 were derived for each of the 15 domains, with higher scores representing greater functioning, greater HRQoL, or greater level of symptoms. Time to deterioration (calculated using the Kaplan-Meier technique) was defined as time from randomization until the date of first clinically meaningful deterioration (a decrease in score from baseline of ≥10) that is confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration.
Time Frame: At baseline, Weeks 3, 6, 9, 12, 16 and 20, then Q4W until PD, on Day 28 and 2 months post-PD, then every 8 weeks until second progression/death (whichever comes first). Assessed until China cohort second analysis DCO (maximum of approximately 29 months).
Population: The China FAS included all randomized patients in the China cohort. For QLQ-C30 function scales and global health status/HRQoL, only patients with baseline scores ≥10 (and with data available) were included in the analysis. For QLQ-C30 symptom scales/items, only patients with baseline scores ≤90 (and with data available) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
months
  QLQ-C30 Global Health Status / HRQoL: number analyzed (Participants) | 60 | 57 | 55
  QLQ-C30 Global Health Status / HRQoL | 14.5 [6.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 15.1 [7.6 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 7.8 [6.5 to 10.9]
  QLQ-C30 Cognitive Functioning: number analyzed (Participants) | 60 | 58 | 58
  QLQ-C30 Cognitive Functioning | 7.6 [4.9 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 6.8 [2.3 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 6.9 [5.7 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  QLQ-C30 Emotional Functioning: number analyzed (Participants) | 60 | 58 | 58
  QLQ-C30 Emotional Functioning | 20.4 [6.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 15.5 [5.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 10.0 [6.9 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  QLQ-C30 Physical Functioning: number analyzed (Participants) | 60 | 58 | 58
  QLQ-C30 Physical Functioning | 21.8 [6.0 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 9.3 [5.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 7.3 [5.7 to 10.9]
  QLQ-C30 Role Functioning: number analyzed (Participants) | 60 | 56 | 57
  QLQ-C30 Role Functioning | 6.8 [4.9 to 21.3] | 6.4 [4.2 to 13.9] | 6.2 [4.1 to 10.0]
  QLQ-C30 Social Functioning: number analyzed (Participants) | 60 | 57 | 56
  QLQ-C30 Social Functioning | 6.7 [4.3 to 14.1] | 5.8 [3.9 to 13.3] | 6.5 [3.3 to 8.3]
  QLQ-C30 Fatigue: number analyzed (Participants) | 60 | 58 | 58
  QLQ-C30 Fatigue | 3.7 [2.3 to 6.8] | 5.3 [2.9 to 9.6] | 3.9 [2.2 to 5.9]
  QLQ-C30 Nausea / Vomiting: number analyzed (Participants) | 59 | 58 | 58
  QLQ-C30 Nausea / Vomiting | 8.4 [4.7 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 9.3 [3.9 to 15.5] | 8.2 [5.7 to 10.9]
  QLQ-C30 Pain: number analyzed (Participants) | 60 | 57 | 58
  QLQ-C30 Pain | 6.6 [4.9 to 17.3] | 6.2 [5.5 to 15.1] | 6.5 [4.6 to 8.6]
  QLQ-C30 Appetite Loss: number analyzed (Participants) | 59 | 57 | 57
  QLQ-C30 Appetite Loss | 8.4 [2.6 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 5.8 [3.3 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 6.9 [5.7 to 10.0]
  QLQ-C30 Constipation: number analyzed (Participants) | 59 | 58 | 58
  QLQ-C30 Constipation | NA [6.8 to NA] — Median and upper limit of 95% CI could not be calculated as they were not reached. | 12.0 [5.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 10.9 [8.6 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  QLQ-C30 Diarrhea: number analyzed (Participants) | 59 | 58 | 58
  QLQ-C30 Diarrhea | 17.3 [9.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | NA [13.3 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 10.1 [8.2 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  QLQ-C30 Dyspnea: number analyzed (Participants) | 60 | 57 | 56
  QLQ-C30 Dyspnea | 11.6 [6.0 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 15.5 [9.3 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 7.3 [5.7 to 10.9]
  QLQ-C30 Insomnia: number analyzed (Participants) | 60 | 57 | 58
  QLQ-C30 Insomnia | 7.3 [5.2 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 15.5 [5.6 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 7.8 [6.3 to 10.9]

30. Secondary Outcome: Time to Deterioration of PRO Symptoms, Assessed Using EORTC QLQ-LC13 in the China Cohort
Description: as for outcome 16
Time Frame: as for outcome 29
Population: The China FAS included all randomized patients in the China cohort. For QLQ-L13 symptom scales/items, only patients with baseline scores ≤90 (and with data available) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 61 | 62
months
  QLQ-LC13 Coughing: number analyzed (Participants) | 58 | 56 | 54
  QLQ-LC13 Coughing | NA [6.8 to NA] — Median and upper limit of 95% CI could not be calculated as they were not reached. | 15.5 [5.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 8.6 [6.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  QLQ-LC13 Dyspnea: number analyzed (Participants) | 60 | 58 | 58
  QLQ-LC13 Dyspnea | 6.9 [3.4 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 8.1 [5.3 to 15.5] | 4.7 [2.5 to 8.6]
  QLQ-LC13 Hemoptysis: number analyzed (Participants) | 60 | 58 | 58
  QLQ-LC13 Hemoptysis | NA [17.3 to NA] — Median and upper limit of 95% CI could not be calculated as they were not reached. | NA [11.2 to NA] — Median and upper limit of 95% CI could not be calculated as they were not reached. | 10.1 [6.9 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  QLQ-LC13 Pain in Arm or Shoulder: number analyzed (Participants) | 60 | 55 | 58
  QLQ-LC13 Pain in Arm or Shoulder | NA [6.9 to NA] — Median and upper limit of 95% CI could not be calculated as they were not reached. | 15.5 [5.6 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 8.6 [6.3 to 10.9]
  QLQ-LC13 Pain in Chest: number analyzed (Participants) | 59 | 55 | 57
  QLQ-LC13 Pain in Chest | NA [6.8 to NA] — Median and upper limit of 95% CI could not be calculated as they were not reached. | 15.5 [6.8 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 10.0 [6.9 to NA] — Upper limit of 95% CI could not be calculated as it was not reached.
  QLQ-LC13 Pain in Other Parts: number analyzed (Participants) | 60 | 58 | 57
  QLQ-LC13 Pain in Other Parts | NA [7.0 to NA] — Median and upper limit of 95% CI could not be calculated as they were not reached. | 9.3 [6.2 to NA] — Upper limit of 95% CI could not be calculated as it was not reached. | 8.6 [5.7 to 10.9]

31. Secondary Outcome: Change From Baseline in Primary PRO Symptoms, Assessed Using EORTC QLQ-C30 and EORTC QLQ-LC13 in the China Cohort; D + T + EP Compared With EP
Description: A MMRM analysis of EORTC QLQ-C30 and EORTC QLQ-LC13 was performed for 5 primary PRO symptoms (cough, dyspnea, chest pain, fatigue and appetite loss), and considered all data from baseline to PD or 12 months, excluding visits with excessive missing data (defined as >75% missing data). An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items, with higher scores representing greater symptom severity. An improvement in symptoms was indicated by a negative change from baseline. A positive change from baseline indicated a deterioration of symptoms. A minimum clinically meaningful change was defined as an absolute change from baseline of ≥10. This outcome measure presents change from baseline for primary PRO symptoms (reported as adjusted means) for analysis of D + T + EP vs EP. Analysis of D + EP vs EP is presented in a separate outcome measure.
Time Frame: as for outcome 17
Population: The China FAS included all randomized patients in the China cohort. For each symptom scale, only patients with data available were included in the analysis.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | China Cohort: D + T + EP | China Cohort: EP
Number analyzed (Participants) | 65 | 62
scores on a scale
  EORTC QLQ-LC13 Cough: number analyzed (Participants) | 60 | 56
  EORTC QLQ-LC13 Cough | -12.8 (2.49) | -12.9 (2.50)
  EORTC QLQ-LC13 Dyspnea: number analyzed (Participants) | 60 | 56
  EORTC QLQ-LC13 Dyspnea | -3.6 (2.21) | -0.8 (2.17)
  EORTC QLQ-LC13 Chest pain: number analyzed (Participants) | 60 | 56
  EORTC QLQ-LC13 Chest pain | -5.1 (2.16) | -5.4 (2.16)
  EORTC QLQ-C30 Fatigue: number analyzed (Participants) | 60 | 56
  EORTC QLQ-C30 Fatigue | 2.8 (2.10) | 2.9 (2.11)
  EORTC QLQ-C30 Appetite loss: number analyzed (Participants) | 60 | 56
  EORTC QLQ-C30 Appetite loss | 3.0 (2.36) | 0.8 (2.42)

32. Secondary Outcome: Change From Baseline in Primary Symptoms as Assessed by EORTC QLQ in the China Cohort; D + EP Compared With EP
Description: as for outcome 18
Time Frame: as for outcome 17
Population: as for outcome 31
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | China Cohort: D + EP | China Cohort: EP
Number analyzed (Participants) | 61 | 62
scores on a scale
  EORTC QLQ-LC13 Cough: number analyzed (Participants) | 58 | 56
  EORTC QLQ-LC13 Cough | -14.9 (2.66) | -16.7 (2.68)
  EORTC QLQ-LC13 Dyspnea: number analyzed (Participants) | 58 | 56
  EORTC QLQ-LC13 Dyspnea | -2.2 (1.93) | -3.0 (1.97)
  EORTC QLQ-LC13 Chest pain: number analyzed (Participants) | 58 | 56
  EORTC QLQ-LC13 Chest pain | -6.7 (1.93) | -7.7 (1.95)
  EORTC QLQ-C30 Fatigue: number analyzed (Participants) | 58 | 56
  EORTC QLQ-C30 Fatigue | 1.5 (2.06) | 0.8 (2.11)
  EORTC QLQ-C30 Appetite loss: number analyzed (Participants) | 58 | 56
  EORTC QLQ-C30 Appetite loss | 3.6 (2.47) | -2.2 (2.51)

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events (TEAEs) were collected up to the final analysis DCO for each cohort; maximum of approximately 33 months for the Global cohort and maximum of approximately 29 months for the China cohort. Serious AEs and Deaths were collected through LTFU analysis in patients still receiving durvalumab (or within 90 days of discontinuing treatment); up to approximately 4 years.
Description: TEAEs included those from first administration of study treatment up to and including 90 days after last dose of study treatment or up to date of initiation of the first subsequent anticancer therapy (whichever occurred first). Data from the global cohort and China cohort safety analysis sets was summarised separately. 6 patients in the China cohort were also included in the global cohort.
Arm/Group | Global Cohort: D + T + EP | Global Cohort: D + EP | Global Cohort: EP | China Cohort: D + T + EP | China Cohort: D + EP | China Cohort: EP
All-Cause Mortality (participants affected / at risk) | 225/266 | 218/265 | 247/266 | 50/65 | 51/61 | 55/62
Serious Adverse Events (participants affected / at risk) | 126/266 | 86/265 | 97/266 | 31/65 | 26/61 | 22/62
Other Adverse Events (participants affected / at risk) | 249/266 | 247/265 | 248/266 | 65/65 | 61/61 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort: D + T + EP (N=266) | Global Cohort: D + EP (N=265) | Global Cohort: EP (N=266) | China Cohort: D + T + EP (N=65) | China Cohort: D + EP (N=61) | China Cohort: EP (N=62)
Anaemia (Blood and lymphatic system disorders) | 9 (11) | 5 (8) | 12 (14) | 2 (2) | 0 (0) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (6) | 7 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (12) | 12 (15) | 12 (13) | 2 (3) | 0 (0) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 7 (12) | 0 (0) | 1 (1) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 2 (3) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 9 (11) | 3 (3) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial prostatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 16 (17) | 6 (6) | 11 (12) | 9 (9) | 5 (5) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza B virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal artery thrombosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort: D + T + EP (N=266) | Global Cohort: D + EP (N=265) | Global Cohort: EP (N=266) | China Cohort: D + T + EP (N=65) | China Cohort: D + EP (N=61) | China Cohort: EP (N=62)
Diarrhoea (Gastrointestinal disorders) | 40 (54) | 27 (37) | 29 (34) | 16 (26) | 5 (5) | 5 (5)
Asthenia (General disorders) | 37 (47) | 42 (50) | 39 (50) | 10 (11) | 6 (8) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 94 (115) | 97 (110) | 116 (150) | 47 (79) | 44 (58) | 44 (62)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 4 (9) | 4 (12)
Leukocytosis (Blood and lymphatic system disorders) | 3 (5) | 4 (4) | 6 (6) | 5 (5) | 2 (2) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 33 (69) | 40 (87) | 32 (69) | 28 (73) | 31 (65) | 22 (69)
Lymphopenia (Blood and lymphatic system disorders) | 8 (12) | 5 (10) | 8 (13) | 6 (11) | 1 (1) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 112 (213) | 110 (221) | 119 (234) | 26 (50) | 22 (40) | 19 (55)
Thrombocytopenia (Blood and lymphatic system disorders) | 50 (68) | 41 (63) | 48 (83) | 15 (28) | 13 (25) | 14 (23)
Hyperthyroidism (Endocrine disorders) | 26 (26) | 26 (28) | 1 (1) | 11 (11) | 7 (8) | 1 (1)
Hypothyroidism (Endocrine disorders) | 28 (33) | 25 (26) | 4 (4) | 13 (14) | 7 (7) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 18 (21) | 14 (16) | 7 (8) | 4 (4) | 7 (9) | 0 (0)
Constipation (Gastrointestinal disorders) | 54 (65) | 43 (53) | 52 (71) | 25 (39) | 24 (29) | 22 (29)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (6) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 85 (126) | 89 (147) | 88 (140) | 31 (72) | 20 (51) | 27 (59)
Stomatitis (Gastrointestinal disorders) | 21 (23) | 8 (10) | 8 (9) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 36 (44) | 39 (65) | 42 (56) | 30 (62) | 19 (35) | 23 (57)
Fatigue (General disorders) | 53 (61) | 48 (61) | 46 (55) | 6 (7) | 7 (7) | 6 (8)
Malaise (General disorders) | 11 (11) | 7 (8) | 3 (3) | 7 (7) | 6 (7) | 4 (6)
Non-cardiac chest pain (General disorders) | 10 (14) | 14 (17) | 7 (8) | 2 (3) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 12 (15) | 16 (19) | 9 (10) | 3 (7) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 36 (53) | 22 (24) | 16 (18) | 23 (33) | 6 (9) | 5 (8)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (7) | 1 (1) | 0 (0) | 10 (12) | 4 (8) | 2 (3)
Nasopharyngitis (Infections and infestations) | 6 (8) | 10 (13) | 7 (8) | 7 (8) | 2 (2) | 3 (3)
Pneumonia (Infections and infestations) | 13 (13) | 8 (10) | 13 (13) | 5 (7) | 3 (4) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 17 (18) | 5 (6) | 7 (7) | 12 (19) | 2 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 8 (10) | 12 (16) | 11 (13) | 4 (5) | 4 (7) | 3 (4)
Alanine aminotransferase increased (Investigations) | 20 (25) | 16 (21) | 12 (15) | 17 (24) | 6 (6) | 6 (10)
Amylase increased (Investigations) | 6 (7) | 11 (12) | 2 (2) | 4 (5) | 4 (8) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (22) | 16 (21) | 9 (11) | 11 (12) | 11 (13) | 5 (7)
Blood alkaline phosphatase increased (Investigations) | 11 (12) | 13 (17) | 6 (7) | 2 (3) | 2 (2) | 4 (4)
Blood bilirubin increased (Investigations) | 5 (5) | 3 (5) | 4 (5) | 7 (12) | 3 (4) | 3 (6)
Blood creatinine increased (Investigations) | 3 (3) | 5 (5) | 6 (6) | 6 (9) | 5 (9) | 5 (8)
Blood lactate dehydrogenase increased (Investigations) | 4 (5) | 6 (6) | 8 (8) | 2 (3) | 1 (3) | 5 (10)
Blood urea increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 2 (2) | 4 (8)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 9 (10) | 13 (13) | 6 (7) | 4 (6) | 2 (3) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 4 (4)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 4 (7) | 3 (8)
Neutrophil count decreased (Investigations) | 11 (16) | 26 (42) | 31 (49) | 22 (52) | 28 (44) | 21 (71)
Platelet count decreased (Investigations) | 6 (8) | 16 (20) | 14 (22) | 10 (15) | 10 (11) | 11 (17)
Weight decreased (Investigations) | 19 (20) | 10 (10) | 9 (10) | 7 (8) | 10 (12) | 5 (6)
White blood cell count decreased (Investigations) | 9 (11) | 14 (21) | 17 (22) | 16 (34) | 17 (27) | 24 (54)
Decreased appetite (Metabolism and nutrition disorders) | 57 (64) | 48 (60) | 46 (54) | 27 (40) | 27 (46) | 27 (54)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (9) | 10 (14) | 9 (11) | 1 (1) | 4 (5) | 3 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (10) | 5 (10) | 7 (9) | 2 (5) | 4 (5) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3) | 4 (4) | 1 (1) | 4 (6) | 3 (10) | 6 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (14) | 5 (6) | 5 (8) | 7 (7) | 3 (4) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (6) | 7 (7) | 2 (2) | 2 (2) | 4 (6)
Hypochloraemia (Metabolism and nutrition disorders) | 5 (6) | 0 (0) | 0 (0) | 5 (9) | 5 (6) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (22) | 17 (21) | 11 (13) | 9 (18) | 9 (12) | 12 (18)
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 (18) | 18 (20) | 13 (14) | 4 (5) | 1 (1) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 20 (28) | 26 (34) | 9 (11) | 18 (28) | 10 (13) | 16 (20)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (5) | 5 (6) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (33) | 24 (32) | 18 (24) | 3 (4) | 3 (4) | 5 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (11) | 5 (6) | 1 (1) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 12 (16) | 4 (4) | 2 (2) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 15 (20) | 23 (27) | 12 (13) | 6 (7) | 6 (8) | 5 (7)
Headache (Nervous system disorders) | 29 (31) | 17 (19) | 22 (25) | 4 (4) | 4 (6) | 2 (3)
Paraesthesia (Nervous system disorders) | 17 (17) | 18 (19) | 13 (15) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 25 (27) | 23 (28) | 13 (14) | 6 (8) | 6 (8) | 8 (13)
Proteinuria (Renal and urinary disorders) | 3 (8) | 1 (3) | 3 (5) | 14 (22) | 9 (14) | 10 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (32) | 35 (36) | 19 (20) | 11 (13) | 8 (8) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (31) | 32 (36) | 27 (30) | 3 (5) | 4 (4) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 12 (13) | 5 (6) | 2 (2) | 7 (7) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10 (18) | 10 (16) | 9 (20) | 5 (6) | 4 (4) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 10 (11) | 6 (7) | 4 (4) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (11) | 7 (8) | 9 (11) | 6 (7) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 79 (80) | 84 (84) | 92 (94) | 28 (29) | 29 (29) | 27 (27)
Pruritus (Skin and subcutaneous tissue disorders) | 40 (52) | 21 (33) | 10 (10) | 4 (14) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 37 (52) | 16 (20) | 10 (10) | 25 (37) | 12 (16) | 2 (2)
Hypertension (Vascular disorders) | 13 (15) | 16 (25) | 7 (8) | 6 (13) | 7 (12) | 3 (8)

LIMITATIONS AND CAVEATS:
Analysis of the China cohort was performed to evaluate the consistency of efficacy and safety in Chinese patients with the global cohort in order to meet regulatory requirements and was not powered for a formal assessment of statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT03043872/Prot_004.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT03043872/SAP_005.pdf